CLINICAL TRIAL: NCT01160965
Title: Ropivacaine 0.75% Versus Levobupivacaine 0.5% for Conversion of Labour Epidural to Surgical Anaesthesia for Emergency Caesarean Section.
Brief Title: Ropivacaine 0.75% Versus Levobupivacaine 0.5% for Conversion of Labour Epidural
Acronym: RoLe
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Not able provide staff for recruting at present
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Dr Geraldine O'Sullivan (Consultant Anaesthetist), Guy's & St Thomas' NHS Foundation Trust
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Version1.0; 2010-021783-15 (EudraCT Number)
Record Dates: First submitted 2010-07-07; First posted 2010-07-13 (Estimated); Last update posted 2011-12-29 (Estimated); Status verified 2011-12

CONDITIONS: Caesarean Section
Keywords: epidural top-up; emergency Caesarean section
MeSH Terms: interventions — Levobupivacaine; Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 0.5% levobupivacaine (Active Comparator): Participants given 15mls of 0.5% levobupivacaine as the solution for their epidural top-up
  Interventions: Drug: 0.5% levobupivacaine
- 0.75% Rpoivacaine (Active Comparator): Participants given 15mls of 0.75% ropivacaine as the solution for their epidural top-up.
  Interventions: Drug: 0.75% Ropivacaine

INTERVENTIONS:
Drug: 0.5% levobupivacaine — 15mls of a 5mg/ml solution of the local anaesthetic levobupivacaine given via the epidural catheter.
  Other Names: 0.5% Chirocaine
  Arms: 0.5% levobupivacaine
Drug: 0.75% Ropivacaine — 15mls of a 7.5mg/ml solution of the local anaesthetic ropivacaine given via the epidural catheter.
  Arms: 0.75% Rpoivacaine

SUMMARY:
The aim of this trial is to compare the local anaesthetic ropivacaine to local anaesthetic levobupivacaine in converting the standard patient controlled labour epidural to provide anaesthesia for an emergency Caesarean section. This is a technique commonly known as an epidural top-up. The investigators set out to disprove the hypothesis that there is no difference between the 2 local anaesthetics in the time of onset and number of times epidural top-up needs supplementing during surgery.

DETAILED DESCRIPTION:
In a randomised controlled trial involving 45 patients the speed of onset of the effects of 20mls of 0.75% ropivacaine was found to be similar to that of 20mls of 0.5% bupivacaine1. However it was also found to be more efficacious at preventing 'breakthrough' pain and therefore had a lower intra-operative supplementation rate. Unfortunately the study was probably not powered adequately to confirm this finding. Bupivacaine has now largely been replaced in the this field by the less cardio-toxic stereoisomer levobupivacaine. A trial comparing 0.75% ropivacaine to 0.5% levobupivacaine and a lignocaine/adrenaline/fentanyl mixture was conducted in Singapore in 20082. It did not show a clinical difference between any of the agents. Whether the population studied is comparable to that in the UK is doubtful and it was not adequately powered to detect a difference in intra-operative supplementation rate. Local experience has shown ropivacaine 0.75% to provide a block with a rapid onset that has little requirement for supplementation intra-operatively. The need to supplement a local anaesthetic block during surgery means that the mother is experiencing a degree of pain that is unacceptable and we view this as a major consideration in choice of local anaesthetic for an epidural top-up. Whilst speed of onset is important, in that it influences the decision to delivery time of the baby, the evaluation of intraoperative supplementation will be a major focus of this trial.

ELIGIBILITY:
Inclusion Criteria:

Any subject requiring a grade 2 or 3 EmCS on the Hospital Birth Centre, St Thomas' who has:

1. Labour analgesia provided by the standard patient controlled epidural (solution containing 0.1% levobupivacaine and 2mcg/ml fentanyl). That is providing analgesia via the patient controlled epidural analgesia infusion pump without the need for multiple extra boluses of epidural local anaesthetic and or opiates from the anaesthetist on the labour ward..
2. Singleton pregnancy.
3. Established labour, determined by the midwife responsible for the patient (usually by vaginal examination of the cervix).
4. Gestation >36 weeks
5. No complex past medical history according to the judgement of the investigator
6. > 18 years of age
7. EmCS starts between the hours 0800 and 1800.
8. The ability to understand the patient information sheet and willing to provide informed consent.
9. Had a minimal total dose of 50mcg of fentanyl since insertion of epidural

Exclusion Criteria:

1. Pre-eclampsia / Eclampsia
2. Antepartum haemorrhage
3. Any congenital, structural or ischaemic heart disease.
4. Category 1 EmCS.
5. Participation in another therapeutic study in the last 12 weeks. -

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2012-08; Primary Completion 2013-08 (Estimated); Study Completion 2014-08 (Estimated)

PRIMARY OUTCOMES:
Supplementation Rate | During operation (approximately 1 hour )
  The number of times the epidural anaesthetic requires intra-operative supplementation with more study solution or another drug for pain.

SECONDARY OUTCOMES:
Pre-operative supplementation | 10-45mins (top-up to start of surgery)
  If further 5mls of study solution is required to achieve block height suitable for surgery to start.
Pain | During operation (approximately 1 hour)
  Incidence of breakthrough pain and its intensity during the operative phase of the Caesarean section
Conversion Rate | At any point between epidural top-up and end of operation (approximately 90mins from epidural top-up)
  If the epidural anaesthetic needs to be converted to spinal anaesthetic or general anaesthetic as it is not adequate for conduction of a Caesarean section
Side effects | At any point between top-up of epidural and end of operation (approximately 90mins from epidural top-up)
  Occurrence of any of nausea, vomiting, itching and shivering during the specified time period
Blood pressure supplementation rate | At any point from top-up of epidural to end of operation (approximately 90mins from epidural top-up)
  Use of the vasopressor phenylephrine and Hartmannn's solution to be given if mean arterial BP drops greater than 30% below baseline or systolic BP of <100mg Hg.
Patient Satisfaction | Prior to leaving operating theatre (approximatelty 120 minutes from epidural top-up)
  Maternal satisfaction, asked to verbally score from 1-10 their satisfaction with the anaesthetic.
Motor block | prior to top-up and prior to leaving theatre (approximatelty 120 minutes from epidural top-up).
  Scored using the Bromage scoring system asking patient to raise legs and noting how able they are to do this.
Fetal Wellbeing | After delivery (approximately 5-10 minutes from start of surgery)
  Neonatal Apgar scores at 1 and 5 minutes after delivery. pH of umbilical blood following delivery
Onset Time | From administration of epidural top-up (approximately 10-45 minutes)
  The time elapsed between administration of the top-up and onset of anaesthesia suitable for surgery to proceed. Defined as a loss of sensation to cold to T4 dermatomal level.

CONTACTS AND LOCATIONS:
Overall Officials: geraldine e o'sullivan, MBBCh, Study Director — Guy's and St Thomas' NHS Foundation Trust
Locations (1):
- St Thomas' Hospital, London, United Kingdom

REFERENCES:
- [Result] Sanders RD, Mallory S, Lucas DN, Chan T, Yeo S, Yentis SM. Extending low-dose epidural analgesia for emergency Caesarean section using ropivacaine 0.75%. Anaesthesia. 2004 Oct;59(10):988-92. doi: 10.1111/j.1365-2044.2004.03753.x. PMID 15488058
- [Result] Sng BL, Pay LL, Sia AT. Comparison of 2% lignocaine with adrenaline and fentanyl, 0.75% ropivacaine and 0.5% levobupivacaine for extension of epidural analgesia for urgent caesarean section after low dose epidural infusion during labour. Anaesth Intensive Care. 2008 Sep;36(5):659-64. doi: 10.1177/0310057X0803600505. PMID 18853583